CLINICAL TRIAL: NCT03126396
Title: Assessment of Efficacy, Tolerance and Acceptability of Urgo 310 3166 Dressing in the Treatment of Local Venous or Mixed Leg Ulcers
Brief Title: Assessment of Efficacy & Tolerance of Urgo 310 3166 Dressing in Local Venous or Mixed Leg Ulcers
Acronym: CASSIOPEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-17-02-310 3166
Record Dates: First submitted 2017-04-11; First posted 2017-04-24 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Ulcers, Leg
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urgo 310 3166 dressing (Experimental): Urgo 310 3166 dressing
  Interventions: Device: Urgo 310 3166 dressing

INTERVENTIONS:
Device: Urgo 310 3166 dressing — Experimental: Urgo 310 3166 dressing

SUMMARY:
Assessment of efficacy & tolerance of Urgo 310 3166 dressing in the treatment of local venous or mixed leg ulcers.

DETAILED DESCRIPTION:
Assessment of efficacy, tolerance and acceptability of Urgo 310 3166 dressing in the treatment of local venous or mixed leg ulcers: multicenter trial, conducted in France.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years old who has provided his/her written informed consent
2. Patient who can be monitored by the same investigation team throughout the whole duration of the study
3. Patient who agrees to wear an effective venous compression system every day, associated with the trial dressing
4. Leg ulcer with an Ankle Brachial Pressure Index (ABPI) not less than 0.7 and not more than 1.3
5. Ulcer area between 3 and 20 cm2
6. Ulcer duration between 3 and 18 months,
7. Ulcer presenting a surface wound bed covered with 50% or more by granulation tissue
8. Moderately or heavily exudative ulcers.

Exclusion Criteria:

A. Clinical infection on the wound bed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Efficacy - % of Wound Area Regression (WAR | at week 12
  % of Wound Area Regression (WAR), as a measure of efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- URGO, Chenôve, France

IPD SHARING:
Plan to Share IPD: No